CLINICAL TRIAL: NCT03037138
Title: Use Of Blood Flow Rate Profiling For Postdialysis Washed-Out Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Collaborators: New Jeddah Clinic Hospital (Industry)
Responsible Party: Principal Investigator, Mahmoud Hamada imam, Lecturer of Nephrology in Internal Medicine Department, Benha University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BenhaU
Record Dates: First submitted 2017-01-24; First posted 2017-01-31 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Hemodialysis-Induced Symptom
Keywords: postdialysis washed-out

STUDY DESIGN:
Intervention Model Description: Use of blood flow profiling for prevention of postdialysis washed-out feeling through same group scale before and after profiling
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Washed-out scale after using BFR profiling (Other): Blood flow profiling will be used as intervention for washed-out dialysis patients
  Interventions: Other: Blood flow Rate profiling

INTERVENTIONS:
Other: Blood flow Rate profiling — Blood flow rate profiling during dialysis session

SUMMARY:
Hemodialysis patients frequently complain of postdialysis fatigue and washed-out feeling. The aim of this study is to use blood flow rate (BFR) profiling to mitigate postdialysis washed-out state.

DETAILED DESCRIPTION:
Hemodialysis patients who complain of the postdialysis washed-out state were recruited. blood flow rate was altered to be 350 ml/min in the first hour of the session then decreased by 50 ml/min hourly for the 4-hour dialysis session. blood flow rate profiling was continued for 9 dialysis sessions (21 Days). Patients were asked to grade their washed-out state on a scale from 1 (no washed-out state) to 5 (severe washed-out state) before and after blood flow rate profiling. Paired t=-test and Wilcoxon Signed Ranks Test were used in appropriate context to compare washed out scale before and after together with urea reduction rate and other blood chemistry tests.

ELIGIBILITY:
Inclusion Criteria:

* Hemodialysis Patient
* Postdialysis washed-out complain

Exclusion Criteria:

* schedule-non complaint patients
* Patients with recent blood pressure drug modification

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-11-12 (Actual); Primary Completion 2016-12-05 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
Washed-out Scale | after 9 modified dialysis session (21 dyas from start of study)
  Scale of washed-out degree after dialysis

SECONDARY OUTCOMES:
Urea reduction Rate | after 9 modified dialysis session (21 dyas from start of study)
  change in urea reduction rate after use of blood flow rate profiling

IPD SHARING:
Plan to Share IPD: No